CLINICAL TRIAL: NCT04113304
Title: Pediatric Motivational mHealth Parent Training for Child Disruptive Behaviors
Brief Title: The Parenting Young Children Check-up: Proof-of-Concept Trial
Status: Completed | Type: Observational
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Lucy (Kathleen) McGoron, Ph.D., Assistant Professor (Research), Wayne State University
Other Study IDs: K01MH110600 (NIH)
Record Dates: First submitted 2019-06-27; First posted 2019-10-02 (Actual); Results first posted 2022-03-24 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Disruptive Behavior Disorders
Keywords: Parenting Interventions; Parent Training; Technology-based intervention; Disruptive Behavior Problems; Early Childhood
MeSH Terms: conditions — Attention Deficit and Disruptive Behavior Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Parenting Young Children Check-up (PYCC) — The PYCC intends to motivate parents to learn behavioral parenting strategies to reduce child disruptive behavior.

SUMMARY:
The Parenting Young Children Check-up (PYCC) is a 3-part system for parents of children with Disruptive Behavior Problems (DBPs). First, at a pediatric visit, parents complete a screener for DBPs and, if reported, go through a tablet-based program to receive feedback and learn about the PYCC. Next, parents receive text messages to connect them to further parent training content. Third, parent training content is delivered via a web-based resource, which includes videos to teach parenting skills. In this proof-of-concept trial, the investigators will examine the acceptability of the tablet-based program and motivation of parents to engage in the PYCC and use the web-based resource.

At a pediatric visit, parents will be told about the research opportunity by a staff member before, during, or after their visit. There will be a flier for parents, which will be available for receptionists to include with in-take paperwork. If parents express openness to participating, a research assistant will meet with them, go over the consent form, and let them complete the screener. Parents will complete a demographics questionnaire and the DBP screener. If parents report elevated DBPs, then they will be eligible to further participate. If they are eligible and choose to participate, the research assistant will have them go through the tablet-based program. Next, they will complete a brief questionnaire asking for input on the PYCC. Each of these components will be completed in the Computerized Intervention Authoring System (CIAS). The brief questionnaire is intended to evaluate perceptions of 1) ease of use, 2) usefulness of the information, 3) likability, and 4) intentions to use the PYCC web-based resource. Items will be rated on a 0 (strongly disagree) to 4 (strongly agree) scale. Parents will also verbally answer 6 open-ended interview questions about the program and suggest improvements. Answers will be audio-recorded and transcribed. All participants (whether only completing the screening or both parts of the study) will receive a resource list as well as a list of URLs to access videos on the video-based content on PYCC website. An ID number will need to be entered to use the website and the investigators will track website use.

This data collection is not hypothesis driven. Rather, the intent is to gather mixed methods feedback from parents to shape the PYCC program.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* English speaking
* Parent to a child ages 2-5
* Report their child has elevated disruptive behavior problems on the Eyberg Child Behavior Inventory

Exclusion Criteria:

* Parent reports child has Autism Spectrum Disorder
* Parent reports child has an intellectual disability
* Parent reports child is receiving treatment for Oppositional Defiant Disorder or Attention Deficit Hyperactivity Disorder

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pediatric primary care clinic; parents that report elevated child disruptive behavior problems
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Merrill Palmer Skillman Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Parents went through the brief tablet-based intervention for the Parenting Young Children Check-up
Period: Overall Study
Arm/Group | Intervention
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intervention
Number analyzed (Participants) | 6
Age, Continuous [Mean (Full Range); unit: years] | 27.83 [23 to 35]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 0
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Intentions to Use the Parenting Young Children Check-up Web-based Resource: Quantitative
Description: Two items (created for this project) were used to assess this outcome. Parents were asked their intentions to use the web-based resource (i.e., videos on the website). Items were rated on 5-point Likert scale (0 = Definitely Disagree, 4 = Definitely Agree). To create the final score, the two items were averaged with a possible range from 0-4 with higher scores indicating stronger intentions to use the Parenting Young Children Check-up web-based resource.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 6
score on a scale | 3.25 [2.00 to 4.00]

2. Primary Outcome: Intentions to Use the Parenting Young Children Check-up Web-based Resource: Qualitative
Description: One oral question, asking if parents intent to use the Parenting Young Children Check-up web-based resource, tapped into this outcome. Responses from participants were coded to reflect what percent of parents were interested in using the web-based resource, what percent of parent are not interested in using the web-based resource, and what percent are unsure.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 6
Participants
  Reported intentions to use program | 6
  Did not report intention to use program | 0

3. Secondary Outcome: Perceived Ease of Use of the Parenting Young Children Check-up Program
Description: Five questionnaire items (created for this project) were used to assess this outcome. Parents were asked about perceived ease of use of each part of the program. Each of the 5 items were rated on a 5-point Likert scale (0 = Definitely Disagree, 4 = Definitely Agree); higher scores indicate more perceived ease of use. An average ease of use score was computed by averaging the responses to the 5 items; the possible range was from 0-4 with higher scores indicate more ease of use).
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 6
score on a scale | 3.40 [2.80 to 4.00]

4. Secondary Outcome: Perceived Usefulness of the Parenting Young Children Check-up Program
Description: Seven questionnaire items (created for this project) were used to assess this outcome. Parents were asked about perceived usefulness of each part of the program. Each of the 5 items were rated on a 5-point Likert scale (0 = Definitely Disagree, 4 = Definitely Agree); higher scores indicate more perceived ease of use. An average usefulness score was computed by averaging the responses to the 5 items; the possible range was from 0-4 with higher scores indicate more ease of use).
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 6
score on a scale | 3.52 [3.00 to 4.00]

5. Secondary Outcome: Likeability of the Parenting Young Children Check-up Program
Description: Four questionnaire items (created for this project) tapped into this outcome. Parents were asked about how much they like each part of the program. Items were rated on a 5-point Likert scale (0 = Definitely Disagree, 4 = Definitely Agree); higher score indicated more likability. An average likability score was computed by taking the average of the 4 responses; possible range from 0-4 with higher scores indicate more likability.
Time Frame: Baseline
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Intervention
Number analyzed (Participants) | 6
score on a scale | 3.63 [3.00 to 4.00]

6. Secondary Outcome: Suggestions for Program Improvements
Description: One oral interview question ("Tell me your ideas about how to make the program better?') will tap into this outcome. Responses will be coded for specific suggestions to improve the Parenting Young Children Check-up program.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 6
Participants
  No changes suggested | 2
  Suggested adding captioning to videos | 1
  Suggested giving out a pamphlet for the program | 1
  Suggested having in-person classes | 1
  Suggested changing voice of program narrator | 1

7. Other Pre Specified Outcome: Number of Participants That Use the Web-based Parent Training Resources
Description: All participating parents will have an ID to access web-based parent training resources. The investigators will track to see who makes use of the resources; the frequency of use (n and % of families that use the web-based resource) will be reported.
Time Frame: Between baseline and 3-months after
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention
Number analyzed (Participants) | 6
Participants
  Used web-based resource | 0
  Did not use web-based resource | 6

ADVERSE EVENTS:
Time Frame: Adverse event data were collected through study completion, which took approximately 25 minutes at one time point.
Description: The clinicaltrials.gov definition was used.
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-01-16): https://cdn.clinicaltrials.gov/large-docs/04/NCT04113304/Prot_SAP_ICF_000.pdf